CLINICAL TRIAL: NCT03135756
Title: Transdiagnostic Endophenotypes of Anxiety and Depression
Brief Title: Mechanisms of Anxiety and Depression Study
Status: Completed | Type: Observational
Sponsor: Palo Alto University (Other)
Responsible Party: Principal Investigator, Stacie Warren, Ph.D., Primary Investigator, Palo Alto University
Other Study IDs: 15-003-H
Record Dates: First submitted 2017-04-21; First posted 2017-05-01 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Depression and anxiety symptoms
- Healthy controls

SUMMARY:
Eligible participants will come in for three separate visits in which they will be interviewed, perform a variety of tasks, and undergo a non-invasive MRI scan. The investigators anticipate that (1) participants with anxiety and depression will likely perform differently than the healthy controls on cognitive tasks, (2) participants with anxiety and depression will likely show differences in brain functionality compared to the healthy controls, and (3) depression and anxiety likely share some underlying mechanisms.

DETAILED DESCRIPTION:
In order to determine eligibility, a brief phone screen lasting approximately 15 minutes will be conducted. If participants are eligible, they will be asked to come in for three separate visits. During the first visit, participants will complete questionnaires as well as a structured interview with one of the study's staff members at Palo Alto University in Los Altos. During the second visit, participants would come to Palo Alto University in Los Altos and complete questionnaires as well as a testing session involving various tasks. During the third visit, participants would undergo a non-invasive brain scan in which participants would complete a task as well as various questionnaires at Stanford University in Stanford.

The investigators have flexible hours and can work around participants' schedules! To inquire more about participation, participants can either email the investigators at paloalto.study@gmail.com or call the investigators at (650) 417-2000 ext. 3642

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* Healthy with no medical conditions OR have a history of anxiety and/or depression
* Ability to travel to both Palo Alto University and Stanford University

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The investigators expect to enroll 50 right-handed, English as first language, adults will be recruited from the community through various advertisements. The investigators expect that 25 will be healthy controls and 25 will be a clinical sample exhibiting clinically significant symptoms of anxiety and depression.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2015-03-19 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
Brain imaging | Day 1
  Non-invasive MRI brain scan to see function and structure of brain
Assessment of symptoms and daily functioning | Day 1
  Structured Clinical Interview for DSM-IV, General demographic questionnaires, Penn State Worry Questionnaire, Intolerance of Uncertainty Questionnaire, The Positive and Negative Affect Schedule, Behavioral Inhibition Scale/Behavioral Activation Scale, The NEO Five-Factor Inventory, Mood and Anxiety Symptom Questionnaire, Alcohol Use Disorders Identification Test, Behavioral Regulation Index and Metacognition Index, General temperament Survey, Questionnaire of Mental Imagery, Rumination Reflection Questionnaire, Drug Abuse Screening Test, Childhood Trauma Questionnaire- Factor Structure, Emotion Regulation Questionnaire, Trait Meta-Mood Scale
Cognitive assessment | Day 1
  Objective assessment of cognitive strengths and weaknesses via neuropsychological testing session

CONTACTS AND LOCATIONS:
Overall Officials: Stacie Warren, PhD, Principal Investigator — Palo Alto University
Locations (2):
- United States (2):
  - Palo Alto University, Los Altos, California
  - Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: Undecided